CLINICAL TRIAL: NCT06812663
Title: Assessment of Some Metabolic and Hematological Markers in Women Exposed to in Vitro Fertilization
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Salah Hassan Omar, residdant doctor, Assiut University
Other Study IDs: metabolic and hematologicalIVF
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: In Vitro Fertilization (IVF)
Keywords: metabolic and hematological markers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- IVF women: Women aged 30 years of age and above, presenting with any infertility concern and BMI 18.5-38 kg/m2.

SUMMARY:
Assisted reproductive technologies (ART) represent commonly utilized management strategies for infertility with multifactorial causes (including genetically predisposed diseases). Amongst ART, in vitro fertilization (IVF) is the most popular. IVF treatment may predispose the mother to increased risks and complications during pregnancy, and there may be adverse fetal outcomes. Hormonal therapies, including oral contraceptives, may impair glucose and lipid metabolism, and promote insulin resistance and inflammation.

In vitro fertilization therapy induces weight gain and impairment in glucose, insulin and lipid homeostasis in failed IVF. Improvement of glucose homeostasis, decrease in thyroid profile and increase in lipid profile in clinical pregnancy are likely a pregnancy-related effect.

Hyperglycemic pregnant women were proven to have a high prevalence of caesarean section, preterm delivery, low one-minute Apgar score, respiratory distress syndrome, neonatal jaundice, admission to the neonatal ICU, infants born large for gestational age (LGA), macrosomia.preconception abnormal glucose metabolism may increase the risk of adverse neonatal outcomes in PCOS women. The monitoring and management of preconception glucose homeostasis and IR are essential methods of improving the neonatal outcomes of PCOS women.

Successful implantation and placentation require well-balanced inflammation and immune tolerance. Apart from white blood cells, the role of platelets in the release of mediators that cause local changes in the inflammatory process is very relevant.

Increased levels of CBC inflammation markers may have a negative impact on IVF outcomes among nonobese women with UI.

Successful embryo implantation requires a favorable endometrium, good-quality embryos and delicate coordination between the embryo and endometrium. The tightly controlled inflammatory response in the window of receptivity is essential for successful implantation and growing evidence suggests that chronic inflammation is associated with RIF.

the aim of this study -To explore effects of IVF therapies on metabolic and endocrinal parameters in IVF-conceived pregnancy and its relation to outcome.

2- To investigate whether there could be an association between hematological infammatory markers and in vitro fertilization (IVF) success

DETAILED DESCRIPTION:
Assisted reproductive technologies (ART) represent commonly utilized management strategies for infertility with multifactorial causes (including genetically predisposed diseases). Amongst ART, in vitro fertilization (IVF) is the most popular. IVF treatment may predispose the mother to increased risks and complications during pregnancy, and there may be adverse fetal outcomes. Hormonal therapies, including oral contraceptives, may impair glucose and lipid metabolism, and promote insulin resistance and inflammation.

In vitro fertilization therapy induces weight gain and impairment in glucose, insulin and lipid homeostasis in failed IVF. Improvement of glucose homeostasis, decrease in thyroid profile and increase in lipid profile in clinical pregnancy are likely a pregnancy-related effect.

Hyperglycemic pregnant women were proven to have a high prevalence of caesarean section, preterm delivery, low one-minute Apgar score, respiratory distress syndrome, neonatal jaundice, admission to the neonatal ICU, infants born large for gestational age (LGA), macrosomia.preconception abnormal glucose metabolism may increase the risk of adverse neonatal outcomes in PCOS women. The monitoring and management of preconception glucose homeostasis and IR are essential methods of improving the neonatal outcomes of PCOS women.

Successful implantation and placentation require well-balanced inflammation and immune tolerance. Apart from white blood cells, the role of platelets in the release of mediators that cause local changes in the inflammatory process is very relevant.

Increased levels of CBC inflammation markers may have a negative impact on IVF outcomes among nonobese women with UI.

Successful embryo implantation requires a favorable endometrium, good-quality embryos and delicate coordination between the embryo and endometrium. The tightly controlled inflammatory response in the window of receptivity is essential for successful implantation and growing evidence suggests that chronic inflammation is associated with RIF.

the aim of this study -To explore effects of IVF therapies on metabolic and endocrinal parameters in IVF-conceived pregnancy and its relation to outcome.

2- To investigate whether there could be an association between hematological infammatory markers and in vitro fertilization (IVF) success

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 years of age and above,
* presenting with any infertility concern
* BMI 18.5-38 kg/m2

Exclusion Criteria:

* current or past history of diabetes mellitus, thyroid dysfunction and any other chronic medical condition such as hepatic, renal, respiratory, haematological and cardiovascular disease. Other exclusion criteria included use of any therapy that may affect glucose homeostasis, thyroid and/or lipid profile

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Women aged 30 years of age and above, presenting with any infertility concern and BMI 18.5-38 kg/m2.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolic marker level | 9 month
  change in glucose levels during pregnancy period in IVF women

IPD SHARING:
Plan to Share IPD: Undecided